CLINICAL TRIAL: NCT02210975
Title: An Investigation of Electrical Stimulation on Gastroesophageal Reflux Disease (GERD) in Patients After Sleeve Gastrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: EndoStim Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL4834906814
Record Dates: First submitted 2014-08-04; First posted 2014-08-07 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: GERD; Sleeve Gastrectomy
Keywords: GERD; LES; Sleeve Gastrectomy; Electrical Stimulation Therapy
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Electrical Stimulation Therapy (Experimental)
  Interventions: Device: LES-Stimulation Device

INTERVENTIONS:
Device: LES-Stimulation Device
  Other Names: EndoStim b.v.

SUMMARY:
Sleeve gastrectomy (SG) has gained popularity as both a staged and a definitive procedure for morbid obesity due to its technical simplicity, low-morbidity and excellent results both for weight loss and control of metabolic syndrome. There are however reports of SG worsening pre-existing GERD or causing new-onset GERD. Because of this, patients with pre-existing GERD have been denied the benefits of SG. In addition, patients that develop post-op GERD cannot undergo traditional anti-reflux surgery since the gastric fundus that is required for fundoplication is removed during the SG. Hence, patients with post-SG GERD not adequately controlled with medication can only opt for the more invasive gastric bypass procedure as their only surgical treatment option.

In a recently reported case study, an obese patient with severe GERD successfully treated with EndoStim underwent SG and maintained adequate GERD control with continued use of LES stimulation therapy. However electrical stimulation was not yet tested systematically in patients with prior gastric operation such as sleeve gastrectomy.

This study will test the hypothesis that electrical stimulation is effective in control of GERD associated with SG.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between 18 - 80 years of age.
2. Subject underwent a sleeve gastrectomy minimum one year prior to enrollment (in order to have reached a stable weight loss plateau).
3. Subject has a history of heartburn, regurgitation or both for >6 month prompting physician recommendation of continual daily use of PPI after sleeve gastrectomy.
4. Baseline off-PPI GERD-HRQL score ≥ 20 following 10-14 days off PPI
5. Baseline off-PPI GERD-HRQLscore is at least 5 points higher than the on-PPI score or a positive relationship between the occurrence of their primary symptom during the pH impedance monitoring (symptom association probability ≥ 95% or a SI score ≥ 50%) is present.
6. Subject who are on standard medical therapy for 6 months or longer and experience discomfort or who are otherwise dissatisfied with GERD symptoms.
7. Subjects with a GERD condition that in the opinion of the PI justifies a minimally invasive reversible procedure prior to attempting a more drastic procedure such as a gastric bypass.
8. Subject has exhibited excessive lower esophageal acid exposure during 24-hour pH-metry of antisecretory therapy performed within 6 months of screening visit; pH < 4 for > 6% of total time.
9. Subject has a resting LES end expiratory pressure ≥ 5mmHg on manometry performed within 6 months of enrollment.
10. Subject has no esophagitis or esophagitis ≤ Grade C (LA classification) on upper endoscopy within 6 months of enrollment.
11. Subject has esophageal body contraction amplitude > 30 mmHg for >30% of swallows and > 30% peristaltic contractions on manometry.
12. Subject has signed the informed consent form and is able to adhere to study visit schedule.

Exclusion Criteria:

1. Subject has any non-GERD esophageal motility disorders.
2. Subject has evidence of obstruction or stricture in the gastric sleeve by a barium swallow and endoscopy.
3. Subject has any significant multisystem diseases.
4. Subject has an autoimmune or a connective tissue disorder (e.g. scleroderma, dematomyositis, Calcinosis-Raynaud's-Esophagus Sclerodactyly Syndrome (CREST), Sjogren's Syndrome, Sharp's Syndrome) requiring therapy in the preceding 2 years.
5. Subject has Barrett's epithelium (> M2; >C1) or any grade of dysplasia.
6. Subject has a hiatal hernia larger than 3 cm.
7. Subject has a body mass index (BMI) greater than 35 kg/m2.
8. Subject has Type 1 Diabetes Mellitus
9. Subject has uncontrolled Type 2 Diabetes Mellitus (T2DM) defined as HbA1c >9.5 in the previous 6 months, or has T2DM for > 10 years.
10. Subject has a history of suspected or confirmed esophageal or gastric cancer.
11. Subject has esophageal or gastric varices.
12. Subject has significant cardiac arrhythmia or ectopy or significant cardiovascular disease.
13. Subject has an existing implanted electrical stimulator (e.g., pacemaker, AICD).
14. Subject requires chronic anticoagulant therapy.
15. Subject has dysphagia or esophageal peptic stricture, excluding Schatzki's ring.
16. Subject of child-bearing potential who is pregnant or intends to become pregnant during the trial period.
17. Subject is currently enrolled in other potentially confounding research.
18. History of any malignancy in the last 2 years.
19. Subject has any condition that, at the discretion of the investigator, would preclude participation in the trial.
20. Weight change of +/- 10% of the EWL (Excess Weight Loss) in the 3 months prior to enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-01 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of any complications that are associated with the investigational stimulation device throughout the follow-up period. | up to 12 month follow-up
Efficacy - Disease specific quality of life | Baseline, 6 and 12 month follow up
  The change in patient's GERD-HRQL, where applicable, from baseline (as measured while off PPI) .

SECONDARY OUTCOMES:
pH-monitoring | Baseline, 6 and 12 month FU
  The change in baseline pH values of % 24-hour esophageal pH< 4.0 and number of reflux events >1minute and >5 minute duration with the same on-stimulation pH parameters at 6 months and at 12 months.
Questionnairres, symptom diary | baseline, 6 and 12 month FU
  Change in symptoms frequency and severity at 6 months vs. baseline and at 12 months vs. baseline as measured by patient symptom diary, structured GI questionnaire, and patients quality of life measured by SF-12.
Anti-secretory medication use | Baseline, 6 and 12 month FU
  Change in anti-secretory medication use as evaluated during the two weeks prior to the 6 mo and 12 mo follow up compared to baseline.
HR-manometry | Baseline, 6 and 12 month FU
  Change in LES end expiratory pressure (LESPpre) and the on-stimulation LES end expiratory pressure (LESPpost) at 6 months and 12 months in mmHg.

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands